CLINICAL TRIAL: NCT06334562
Title: An Observational Study on the Clinical Effect of Sugammadex Sodium (Domestic) for Antagonizing Neuromuscular Blockade After Thoracic Surgery
Brief Title: The Clinical Effect of Sugammadex Sodium (Domestic) for Antagonizing Neuromuscular Blockade After Thoracic Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Fourth Affiliated Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KY-2023-112
Record Dates: First submitted 2024-03-14; First posted 2024-03-28 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Neuromuscular Blockade
Keywords: Sugammadex Sodium; Postoperative Neuromuscular Block Antagonism; thoracic surgery
MeSH Terms: interventions — Sugammadex; Neostigmine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sugammadex Sodium group (Experimental): The dose of Sugammadex Sodium is 2mg/kg
  Interventions: Drug: SUGAMMADEX SODIUM 100 Mg in 1 mL
- Neostigmine group (Active Comparator): The dose of Neostigmine is 50 μg/kg
  Interventions: Drug: Neostigmine

INTERVENTIONS:
Drug: SUGAMMADEX SODIUM 100 Mg in 1 mL — The dose of Sugammadex Sodium 100 Mg in 1 mL is 2mg/kg
  Other Names: Sugammadex Sodium
  Arms: Sugammadex Sodium group
Drug: Neostigmine — Neostigmine is 50 μg/kg
  Arms: Neostigmine group

SUMMARY:
This study aims to compare the use of sugammadex (domestic) and neostigmine for antagonism after thoracic surgery, and observe the effect of sugammadex (domestic) on neuromuscular blockade antagonism after thoracic surgery, in order to provide a basis for optimizing the use of muscle relaxants and their antagonists during anesthesia.

DETAILED DESCRIPTION:
All patients were well prepared preoperatively, and vital signs monitoring and accelerated muscle relaxation monitor and TOF monitoring of muscle relaxation were improved after admission. General anaesthesia was induced and maintained by an experienced anaesthesiologist according to the routine drug administration protocol. The neuromuscular blocking drug was limited to rocuronium bromide at an induction dose of 0.6 mg/kg. Anaesthesia was induced with intravenous propofol and maintained with sevoflurane, and rocuronium bromide 0.15 mg/kg. At the end of surgery when the patient's degree of neuromuscular blockade spontaneously recovered to T2 reappearance, the neuromuscular blocking effect of rocuronium bromide was reversed by intravenous rapid injection of sugammadex (domestic) injection or neostigmine within 10 s. The dose of sugammadex (domestic) was 2 mg/kg, and neostigmine 50 μg/kg. Information on dosage and time of neuromuscular blocking medication was recorded, and the patients were recorded at the end of the surgery. Neuromuscular function and clinical performance after reversal with sugammadex (domestic) at the end of the procedure, recording the recovery time of neuromuscular function, extubation time, and time of leaving the room.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who undergo elective lung surgery under general anesthesia and require endotracheal intubation;
2. Age>18 years old, gender not limited;
3. American Society of Anesthesiologists ASA Level I-III;
4. Use rocuronium bromide for neuromuscular blockade;
5. The patient voluntarily participated in the trial.

Exclusion Criteria:

1. The patient explicitly refused to participate in this trial;
2. Family history of malignant hyperthermia, patients with allergies to sodium sulbactam, neostigmine ingredients and their excipients, and patients with allergies to drugs used during general anesthesia;
3. Patients with tracheal malformations or suspected difficult airways, coagulation dysfunction, severe liver and kidney dysfunction, and severe lung disease;
4. Patients who are not extubated and sent to the ward or ICU after surgery;
5. The researchers believe that patients with any other unfavorable factors to participate in this trial.

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Muscle relaxation recovery time | Usually from half an hour to several hours（depending on the length of the procedure）
  The time from using antagonists to TOFr recovery to 0.9

CONTACTS AND LOCATIONS:
Overall Officials: JianHong Xu, Principal Investigator — The Fourth Affiliated Hospital of Zhejiang University School of Medicine
Locations (1):
- The Fourth Affiliated Hospital of Zhejiang University School of Medicine, Yiwu, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No